CLINICAL TRIAL: NCT05629481
Title: a Prospective Single-center, Participant-blinded, Randomized Controlled Clinical Trial of Fractional Carbon Dioxide Laser Treatment for Female Stress Urinary Incontinence
Brief Title: A Study of Fractional Carbon Dioxide Laser Treatment for Female Stress Urinary Incontinence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Yueqing Tang, Principal Investigator, Qilu Hospital of Shandong University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: QL-URO-002
Record Dates: First submitted 2022-11-14; First posted 2022-11-29 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2022-11

CONDITIONS: Stress Urinary Incontinence
Keywords: treatment
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CO2 laser group (Experimental): Participants in the CO2 laser group underwent three vaginal fractional CO2 laser (AcuPulse, Lumenis, Yokneam Illit, Israel) treatment sessions with 4-6 weeks intervals.
  Interventions: Procedure: Fractional carbon dioxide laser treatment
- Sham group (Sham Comparator): Participants in the sham group underwent three sham treatment sessions with 4-6 weeks intervals.
  Interventions: Procedure: Fractional carbon dioxide laser sham treatment

INTERVENTIONS:
Procedure: Fractional carbon dioxide laser treatment — Participants underwent three vaginal fractional CO2 laser (AcuPulse, Lumenis, Yokneam Illit, Israel) treatment sessions with 4-6 weeks intervals. The same laser device parameters (10 mJ, 10% density, spot diameter of 12×12 mm2) were used in participants. A special laser probe was inserted into the patient's vagina after cleaning and disinfection. The laser procedure was performed at the 0, 2, 4, 6, 8, and 10 o'clock positions by rotating the laser probe from the proximal vagina to the distal, and additional procedures were performed at the 11 and 1 o'clock positions 5 mm above the introitus vaginae.
  Arms: CO2 laser group
Procedure: Fractional carbon dioxide laser sham treatment — Participants underwent three vaginal fractional CO2 laser (AcuPulse, Lumenis, Yokneam Illit, Israel) sham treatment sessions with 4-6 weeks intervals. A special laser probe was inserted into the patient's vagina after cleaning and disinfection. The sham procedure was performed at the 0, 2, 4, 6, 8, and 10 o'clock positions by rotating the laser probe from the proximal vagina to the distal, and additional sham procedures were performed at the 11 and 1 o'clock positions 5 mm above the introitus vaginae.
  Arms: Sham group

SUMMARY:
Urinary incontinence (UI) is a common disease that refers to involuntary loss of urine. The prevalence of female UI varies widely across different studies, mostly ranging from 25-40%. Stress urinary incontinence (SUI) is the most common type of UI. SUI is defined as involuntary loss of urine when abdominal pressure increases suddenly such as coughing or sneezing. SUI affects women's quality of life seriously, causing psychological problems such as anxiety and depression, even socialization difficulties. There are many treatment options for female SUI, including non-surgical and surgical interventions. Clinicians and patients need a highly effective and low-risk therapy urgently, thus energy-based therapies were born on demand. This study aims to demonstrate the efficacy and safety of the fractional CO2 laser in the treatment of female SUI, as well as its impact on women's quality of life.

DETAILED DESCRIPTION:
Urinary incontinence (UI) is a common disease that refers to involuntary loss of urine. The prevalence of female UI varies widely across different studies, mostly ranging from 25-40%. Stress urinary incontinence (SUI) is the most common type of UI. SUI is defined as involuntary loss of urine when abdominal pressure increases suddenly such as coughing or sneezing. SUI affects women's quality of life seriously, causing psychological problems such as anxiety and depression, even socialization difficulties.

There are many treatment options for female SUI, including non-surgical and surgical interventions. For example, pelvic floor muscle training (PFMT) is the primary non-surgical treatment method, requiring females to perform Kegel exercises consistently. PMFT has been shown to be effective for female SUI, but the efficacy is dependent on the quality of PMFT. Outpatient PFMT has a higher objective cure rate compared with home PFMT. Surgery is the most effective treatment option, and the most common procedure is the mid-urethral sling (MUS). Nevertheless, surgical risks such as persistent pain after surgery, bleeding, infection, and urinary dysfunction cannot be ignored. Many outpatients are unable to persist in performing high-quality PFMT and do not consent to surgical treatment. Clinicians and patients need a highly effective and low-risk therapy urgently, thus energy-based therapies were born on demand.The result of energy-based therapies including radiofrequency (RF), Erbium: YAG (Er: YAG) laser, and CO2 laser is controversial, which has been reported in several papers. This study aims to demonstrate the efficacy and safety of the fractional CO2 laser in the treatment of female SUI, as well as its impact on women's quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-70 years
* Clinical diagnosis of stress urinary incontinence (SUI)

Exclusion Criteria:

* pregnancy
* pelvic organs prolapse no more than grade II
* gynecologic and urinary tract infections
* previous surgical intervention for stress urinary incontinence (SUI)
* Urgency urinary incontinence (UUI) or Mixed urinary incontinence (MUI)
* serious chronic disease or other reasons that compromised safety and interfered with study compliance

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-04-20 (Actual); Primary Completion 2023-04-20 (Estimated); Study Completion 2023-04-20 (Estimated)

PRIMARY OUTCOMES:
treatment efficacy | through study completion, an average of 6 months
  1-hour pad test, used to assess improvement in the amount of urine leakage. That pad weight increases >2g is considered positive. The improvement criteria was considered as 1-h pad test weight decreasing > 50% baseline.

SECONDARY OUTCOMES:
King's Health Questionnaire (KHQ) score decreases more than 50% baseline | through study completion, an average of 6 months
  King's Health Questionnaire (KHQ) contains 3 parts consisting of 21 items. The subscales in Part 1 and Part 2 scored from 0 to 100. The urinary symptoms scale in Part 3 is scored from 0 to 30. Every subscale and urinary symptoms scale calculate the score respectively and lower scores indicate better quality of life.
Incontinence-specific Quality of Life (I-QOL) score increases more than 50% baseline | through study completion, an average of 6 months
  Incontinence-specific Quality of Life (I-QOL) contains three subscales including avoidance or limiting behaviors (8 items), psychological impacts (9 items), and social embarrassment (5 items). Overall assessment and three subscales of I-QOL scored from 0 to 100, and higher scores indicate better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Zhonghua Xu, MD, Study Chair — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No
Investigators will try to protect the information of the included participants

REFERENCES:
- [Background] Palacios S, Ramirez M. Efficacy of the use of fractional CO2RE intima laser treatment in stress and mixed urinary incontinence. Eur J Obstet Gynecol Reprod Biol. 2020 Jan;244:95-100. doi: 10.1016/j.ejogrb.2019.10.048. Epub 2019 Nov 12. PMID 31778906
- [Result] Alexander JW, Karjalainen P, Ow LL, Kulkarni M, Lee JK, Karjalainen T, Leitch A, Ryan G, Rosamilia A. CO2 surgical laser for treatment of stress urinary incontinence in women: a randomized controlled trial. Am J Obstet Gynecol. 2022 Sep;227(3):473.e1-473.e12. doi: 10.1016/j.ajog.2022.05.054. Epub 2022 May 31. PMID 35662546
- [Result] Amiragova MG, Arakhangel'skaia MI. [Role of the midbrain reticular formation in hormonal supply to the body in conditions of chronic emotional stress]. Biull Eksp Biol Med. 1983 Aug;96(8):16-21. Russian. PMID 6683978
- [Result] Franic D, Fistonic I, Franic-Ivanisevic M, Perdija Z, Krizmaric M. Pixel CO2 Laser for the Treatment of Stress Urinary Incontinence: A Prospective Observational Multicenter Study. Lasers Surg Med. 2021 Apr;53(4):514-520. doi: 10.1002/lsm.23319. Epub 2020 Sep 8. PMID 32896930
- [Result] O'Toole AW, O'Toole R, Webster SW, Lucal B. Nurses' diagnostic work on possible physical child abuse. Public Health Nurs. 1996 Oct;13(5):337-44. doi: 10.1111/j.1525-1446.1996.tb00259.x. PMID 8918174